CLINICAL TRIAL: NCT01703351
Title: Prospective Randomized Trial Comparing the Effectiveness of Continuous Paravertebral Infusion of Local Anesthetics Versus Intravenous Patient-controlled Analgesia on Acute and Chronic Neuropathic Pain After VATS Lobectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2012-0470
Record Dates: First submitted 2012-09-27; First posted 2012-10-10 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Lung Neoplasms; Postoperative Pain
Keywords: pain control, VATS
MeSH Terms: conditions — Lung Neoplasms; Pain, Postoperative; Agnosia | interventions — Ropivacaine; Fentanyl; Nefopam; ramosetron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug: 0.5% ropivacaine (Experimental)
  Interventions: Drug: 0.5% ropivacaine
- Fentanyl 500mcg + acupan 160mg + nasea 0.6mg (Active Comparator)
  Interventions: Drug: Fentanyl 500mcg + acupan 160mg + nasea 0.6mg

INTERVENTIONS:
Drug: 0.5% ropivacaine — (n=48); continuous paravertebral infusion of local anesthetics (0.5% ropivacaine, 5cc/hr for 60 hours after operation) thorough catheter below the parietal pleura using On-Q® system(I-flow corp, Lake Forest, CA, USA)
  Arms: Drug: 0.5% ropivacaine
Drug: Fentanyl 500mcg + acupan 160mg + nasea 0.6mg — (n=48); IV PCA (Fentanyl 500mcg + acupan 160mg + nasea 0.6mg, 5cc/hr for 60 hours after operation, 0.5cc bolus if patients feel breakthrough pain)
  Arms: Fentanyl 500mcg + acupan 160mg + nasea 0.6mg

SUMMARY:
Since mid-2000, thoracoscopic lobectomy has been replaced with conventional open lobectomy and it has reduced the operative morbidities and mortalities. However, thoracoscopic lobectomy also results in operative acute pain and the incidence of chronic pain after thoracoscopic lobectomy has been reported as up to 50%. Penetration of chest wall by trocar, torque at trocar and working window by operator, and compression of intercostal nerves have been suggested as a cause of pain after thoracoscopic lobectomy. The intravenous patient-controlled analgesia (IV PCA) that usually have used to control the operative pain, sometimes cause the side effects such as sedation, nausea and vomiting due to its systemic delivery of analgesics. Because of these side effects, IV PCA has to be discontinues and the effective dose of analgesics could not deliver to patients. In contrast to IV PCA, continuous paravertebral infusion of local anesthetics thorough catheter below the parietal pleura might reduce the side effects of IV PCA and control the operative pain effectively. In this study, we investigate the effectiveness of continuous paravertebral infusion of local anesthetics thorough catheter below the parietal pleura for 60 hours after operation competed to IV PCA.

ELIGIBILITY:
Inclusion Criteria:

* Age; 18≥, <75
* Thoracoscopic lobectomy due to lung cancer or suspected lung cancer
* Tolerable cardiopulmonary and other systemic function tolerable to lobectomy
* Karnofsky performance status ≥ 80
* Agree with study

Exclusion Criteria:

* Intolerable to one-lung ventilation
* Bleeding risk due to Aspirin, coumadin and other drugs
* Past or current history of depression or other psychiatric disease
* Pain persisted before operation due to lung lesion
* History of rib fracture, trauma or lung surgery at the same side of operation
* Severe pleural adhesion or empyema
* Open thoracotomy conversion
* Reoperation due to postoperative bleeding or others
* Postoperative complications that need ICU care
* Chemical pleurodesis more than two times after operation
* Do not agree with study

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-10-04; Primary Completion 2015-11-06 (Actual); Study Completion 2015-11-06 (Actual)

PRIMARY OUTCOMES:
1. Acute pain | Pain score(Visual Analogue Scale) measured in operative day, POD #1, #2, #3, #4)

SECONDARY OUTCOMES:
2. Quality of life | measured Quality of life by EORTC QLQ C 30 (V 3.0) in 4, 8, 12 weeks after operation

OTHER OUTCOMES:
3. Neuropathic pain | VAS score and dose of analgesics in 4, 12 weeks after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Thoracic and Cardiovascular Surgery, Yonsei University College of Medicine, Seoul, South Korea